CLINICAL TRIAL: NCT05754359
Title: Feasibility of an Intervention to Promote Physical Activity in Preschool Children: A Cluster Randomised Controlled Trial
Brief Title: Development and Feasibility of an Intervention to Increase Physical Activity Among Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, NeilHeron, Principal Investigator, Neil Heron, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHLS 22_157
Record Dates: First submitted 2023-02-06; First posted 2023-03-03 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Childhood Obesity; Physical Activity
Keywords: Feasibility; Physical activity; Young Children; Intervention,
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I'm an Active Hero (IAAH) Intervention program (intervention group) (Experimental): Preschool where the intervention implement will be run.
  Interventions: Behavioral: I'm an Active Hero (IAAH) Intervention Program
- Usual physical activities (control group) (No Intervention): No intervention will be delivered in the control group, and children were requested to continue their usual physical activities.

INTERVENTIONS:
Behavioral: I'm an Active Hero (IAAH) Intervention Program — The "I'm an Active Hero (IAAH)" programme is a 10-week intervention aimed at increasing physical activity and decreasing sedentary behaviour in preschool-aged (aged 3-5 years) children. It is anticipated to begin in February 2023 to May 2023. Assessments will be conducted at baseline and immediately following the intervention. The IAAH-intervention will be implemented by the preschool teachers, who will have two teacher training sessions with the main researcher (myself). The IAAH-intervention involves environmental modifications (a classroom) to create areas with sufficient space for active play; classroom sessions these will be implemented for 10 weeks (a minimum of one hour per week); and parent involvement, such as the provision of parental-child interaction homework activities and written information (tip cards, posters, and newsletters). for parents on how to encourage their children to be active.
  Arms: I'm an Active Hero (IAAH) Intervention program (intervention group)

SUMMARY:
The aim of this study is to develop, implement, and evaluate a novel intervention to increase physical activity and reduce sedentary behaviour among pre-school children, with the ultimate goal of reducing obesity among this age group. This study will provide evidence-based recommendations for reducing the prevalence of obesity among preschool-aged children, and the suggestions will help improve the physical activity intervention programme in preschoolers.

DETAILED DESCRIPTION:
The pre-school-based I'm an Active Hero (IAAH) intervention with family involvement was developed in accordance with the Medical Research Council (MRC) framework for developing and evaluating complex interventions. The development phase consists of locating and synthesising existing evidence (such as what is already known about existing interventions) and finding and developing theories (e.g., developing a theoretical understanding of the expected process of behaviour change). The IAAH-intervention components are theory- and evidence-based; they were developed based on a comprehensive identification and evaluation of current and past community, preschool, and family-based physical activity and lifestyle change interventions, as well as recommendations from a recent systematic review and review of reviews.

Additionally, the IAAH-intervention component was informed by conducting a systematic review to identify promising intervention components, including behaviour change techniques, that are associated with interventions that were able to increase PA in the preschool age group. In addition to conducting a qualitative study with teachers and patients/guardians, investigators will also consult them on the intervention's content and duration. Investigators would consider the suggestions and ideas from the preschool practitioners' and parent/guardian focus group meetings, which will establish the meaning of PA for the two distinct stakeholder groups, their influences on this, and considerations for a future intervention. The Template for Intervention Description and Replication (TIDieR) framework was also used to set up the intervention component.

The design of the intervention will employ systematic review and qualitative phases to inform the quantitative, feasibility phase, followed by a further qualitative phase (stakeholders will be involved in the further refinement of the intervention to add richness and depth). Findings from the systematic review and qualitative work will inform the development of the IAAH intervention.

Intervention: This will be a feasibility study of a two-arm cluster-randomised controlled trial (RCT) and will consist of an intervention group and a control group with two data collection time points (i.e., baseline and post-intervention) to test the feasibility and efficacy of a 10-week "I'm an Active Hero (IAAH)" programme intervention with the aim of improving physical activity and decreasing sedentary behaviour of preschool children aged between 3 and 5 years in Taif City, Saudi Arabia.

Process evaluation: This will be a qualitative study including interviews and/or questionnaires with stakeholders (pre-school principals, teachers, classroom assistants, and parents/guardians) to determine the acceptability of the intervention from the participants' perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Children in the preschool years, ages 3 to 5, whose parents or guardians consent to their participation in the study
* An ambulatory individual who does not require physical assistance
* Children who able to follow verbal instructions

Exclusion Criteria:

* Children older than 5 years old
* Children for whom parental/caregiver consent is not provided
* Children with a concurrent medical condition that affects their ability to physically walk a certain distance or with health issues that might influence their participation in the intervention

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Preschool Facilities that Agreed to Participate | 10 weeks
  The proportion of preschools that agreed to take part in the study.(Outcome related to trial feasibility)
Preschool Retention | 10 weeks post baseline
  The percentage of preschools which were retained throughout the study.(Outcome related to trial feasibility)
Participant Recruitment | 10 weeks
  The expected number of participants to be recruited in this study. (Outcome related to trial feasibility).
Participants Retention | 10 weeks post baseline
  The proportion of participants who will complete outcome assessments In either (intervention and control group).(Outcome related to trial feasibility).
Baseline Week ActiGraph Accelerometers-GT3X Return Rate at the End of the Baseline Week | 1 week
  Number of children who will return their ActiGraph accelerometers-GT3X at the end of baseline week on the scheduled day (all children wore the accelerometers simultaneously)
Return of ActiGraph Accelerometers-GT3X on Time by Post-baseline Week Participants | 10 weeks after baseline
  The number of participants who will return their ActiGraph accelerometers-GT3X to the researcher on the designated day, at end of post-baseline week.
Damaged or Lost ActiGraph Accelerometers-GT3X | 11 weeks (1 week at baseline and 10 weeks after baseline
  Number of ActiGraph accelerometers-GT3X that may loss or damage during this study
Intervention Fidelity | 10 weeks
  Intervention fidelity will be undertaken using the teacher's logbook of the number of sessions conducted per week and structure followed in relation to classroom guides) and observing the delivery of interventions, including two sessions of physical activity and sedentary behaviour will be observed at intervention pre-school at the midpoint through the intervention. At the end of the intervention, teachers and parents will be asked to take part in focus group and /or questionnaires.(Outcome related to trial feasibility).
Acceptability : Intervention Acceptance | 1 week after the end of the intervention
  Intervention acceptance will be assessed via a post-intervention acceptance questionnaire and/or qualitative data from a post-intervention focus group.(outcome related to trial acceptability).

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI z-score) Measurement | Baseline and 10 weeks post-intervention
  Height (to 0.1cm) and weight (to 0.1kg) will be measured twice without socks or shoes, in indoor clothing. BMI will then derive, and z -scores created relative to UK1990 data.
Change in Participants Physical Activity from Baseline to Post-intervention | Baseline and 10 weeks post-intervention
  The children's preschool and home physical activity will be monitored objectively using the ActiGraph accelerometers-GT3X to be worn for four consecutive days at baseline and again for four consecutive days in week 11 of the trial. The unit of measurement will be the daily mean of time spent in light, and moderate-vigorous physical activity (LMVPA).
Change in Participants Sedentary Behaviour from Baseline to Post-intervention | Baseline and 10 weeks post-intervention
  The children's preschool and home sedentary behaviour will be measured objectively using the ActiGraph accelerometers-GT3X to be worn at baseline for Four consecutive days and in week 11 of the study again for four consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Neil Heron, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- General Administration of Education in Taif-KSA, Ta'if, Maccha, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Walah MA, Donnelly M, Alhusaini AA, Heron N. Pre-school-based behaviour change intervention to increase physical activity levels amongst young children: a feasibility cluster randomised controlled trial. Front Public Health. 2024 May 2;12:1379582. doi: 10.3389/fpubh.2024.1379582. eCollection 2024. PMID 38756888